CLINICAL TRIAL: NCT02803450
Title: Epidural Loading With High Volume, Low Concentration Prior to Catheter Insertion: is How You Administer the Volume Important?
Brief Title: Epidural Loading: High Volume, Low Concentration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol will be rewritten.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Goran Ristev, Assistant Clinical Professor of Anesthesiology, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2013H0188
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Labor and Delivery
Keywords: Effects of; Anesthesia; spinal and epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Volume, Low Concentration via Epidural Needle (Experimental): Epidural loading: Participants will receive 20ml of 0.0625% bupivacaine with fentanyl 1mcg/ml epidural loading dose in 10ml increments five minutes apart via epidural needle followed by catheter placement.
  For continuous infusions: The continuous patient controlled epidural anesthesia (PCEA) pump will contain 0.03125% bupivacaine with 1mcg/ml fentanyl. The infusion rate will be set at 20ml/hr basal rate and 8ml every 15 minutes on demand with lockout of 52ml/hr.
  For inadequate analgesia: One additional 10ml boluses of the experimental 0.0625% bupivacaine with 1mcg/ml will be provided spaced 5 minutes apart via the epidural catheter.
  Interventions: Procedure: Epidural needle
- High Volume, Low Concentration via Epidural Catheter (Experimental): Epidural loading: Participants will receive 20ml of 0.0625% bupivacaine with fentanyl 1mcg/ml epidural loading dose in 10ml increments five minutes apart via the epidural catheter administration following catheter placement.
  For continuous infusions: The continuous patient controlled epidural anesthesia (PCEA) pump will contain 0.03125% bupivacaine with 1mcg/ml fentanyl. The infusion rate will be set at 20ml/hr basal rate and 8ml every 15 minutes on demand with lockout of 52ml/hr.
  For inadequate analgesia: One additional 10ml boluses of the experimental 0.0625% bupivacaine with 1mcg/ml will be provided spaced 5 minutes apart via the epidural catheter.
  Interventions: Procedure: Catheter Administration
- Low Volume, High Concentration via Epidural Catheter (Active Comparator): Standard of Care Epidural Administration Epidural loading: Participants will receive 10ml of 0.125% bupivacaine with fentanyl 2mcg/ml in 5 ml increments 5 minutes apart via the epidural catheter following epidural catheter placement, per standard of care.
  For continuous infusions: The continuous patient controlled epidural anesthesia (PCEA) pump will contain 0.0625% bupivacaine with 2mcg/ml fentanyl. The infusion rate will be set at 10ml/hr basal rate and 4ml every 15 minutes on demand with lockout of 26ml/hr.
  For inadequate analgesia: One additional 5ml boluses of the standard 0.125% bupivacaine with 2mcg/ml will be provided spaced 5 minutes apart via the epidural catheter.
  Interventions: Procedure: Standard of Care Epidural Administration

INTERVENTIONS:
Procedure: Epidural needle — Medication administration via epidural needle.
  Arms: High Volume, Low Concentration via Epidural Needle
Procedure: Catheter Administration — Medication administration via epidural catheter.
  Arms: High Volume, Low Concentration via Epidural Catheter
Procedure: Standard of Care Epidural Administration — Medication administered at higher concentration, lower volume via epidural catheter.
  Other Names: Epidural catheter
  Arms: Low Volume, High Concentration via Epidural Catheter

SUMMARY:
This prospective, randomized, single blinded control trial will investigate the effects of epidural loading with a high volume, low concentration local anesthetic solution via the epidural needle versus the epidural catheter.

DETAILED DESCRIPTION:
This prospective, randomized, single blinded control trial will investigate the effects of epidural loading with a high volume, low concentration local anesthetic solution via the epidural needle versus the epidural catheter. Control patients will receive local anesthetic in lower volume more concentrated solution via the epidural catheter which is current standard practice. Outcome measures will include quantifying pain relief with respect to time using VAS scores. In addition, post delivery patient satisfaction regarding anesthesia regimen, blood pressure changes, heart rate, anesthetic level, total dose of epidural used during labor, rescue doses and incidence of fetal bradycardia will be assessed. 35 patients will be recruited for each of the three arms of the study, totaling 105 patients, in order to obtain significance when performing statistical analyses following complete enrollment in the study. The impetus of this study involves investigation of the effects of loading the epidural space with high volume, low concentration local anesthetic via two different modalities and studying which method is more efficacious.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have volunteered and consented to participation in the study upon admission to labor and delivery
2. Parturients in active labor requesting epidural analgesia
3. Uncomplicated pregnancy with a reassuring fetal heart tracing
4. Age greater than or equal to 18 years

Exclusion Criteria:

1. Contraindication to epidural anesthesia
2. Inability to read, comprehend, and sign the informed consent form
3. Fetal intrauterine growth retardation (IUGR)
4. Non-reassuring fetal heart tracing
5. Cervical dilation greater than 7cm
6. Intra-uterine fetal demise
7. History of chronic pain other than in the back
8. Incarcerated patients I. Any patient enrolled in the study in whom there is evidence of dural puncture during epidural technique (>3 attempts, presence of CSF)

j. Any evidence of high spinal after initial bolus or continuous infusion of high volume, low concentration local anesthetic solution k. Women undergoing cesarean section

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Patient Pain Levels (VAS Assessment) | During Labor
  Patients will be assessed for pain levels on the VAS scale after analgesia administration in both arms
Patient Satisfaction | During labor
  Patient satisfaction with analgesia using a Likert rating of patient satisfaction with anesthetic care.

SECONDARY OUTCOMES:
Analgesic level | 20 minutes
  Pinprick every 10, 15, and 20 minutes following loading
Maternal Vital Signs | 20 minutes
  Measure change in maternal blood pressure and heart rate over 20 minutes following loading.
Fetal Heart Rate | 20 minutes
  Measure change in fetal heart rate following loading.
Rescue Bolus | During Labor
  Measure number of rescue bolus doses and total anesthetic dose
Intravascular Catheter Placement | During labor
  Measure incidence of intravascular catheter placement.

CONTACTS AND LOCATIONS:
Overall Officials: Goran Ristev, MD, Principal Investigator — The Ohio State Univeristy
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No